CLINICAL TRIAL: NCT06734923
Title: Survey on Media and Social Networks Consultation Among Patients Taken Care in the Orthodontics Unit At the Nice University Hospital: a Cross-sectional Study
Brief Title: Media and Social Networks Consultation and Associated Factors Among Orthodontic Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Odonto03
Record Dates: First submitted 2024-12-05; First posted 2024-12-16 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Dental Care; Using Social Media and Networks to Find Out About Orthodontic Treatment
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient who has conducted online research on orthodontics: online research on orthodontics
  Interventions: Other: Questionnaire (28 questions)

INTERVENTIONS:
Other: Questionnaire (28 questions) — demographic data, information-seeking behavior, platform use and online consultation habits, trust and impact, and interest in additional resources

SUMMARY:
"Context : An increasing number of patients are using the internet and social media to obtain information about oral health, including the field of orthodontics.

Aim : This study aimed to analyze the behavior and habits of patients regarding the use of social media to obtain information about orthodontics, as well as the factors associated with this usage.

Materials and methods : The study was designed as a single-center, cross-sectional, descriptive study. Orthodontic patients filled out a 28-question questionnaire that gathered demographic data, information-seeking behavior, platform use and online consultation habits, trust and impact, and interest in additional resources. A univariate and multivariate logistic regression models/analysis were conducted using Excel and IBM SPSS Statistics Version 29.0.1.0, (employing Chi2, Fisher's exact tests, univariate and multivariate models)."

ELIGIBILITY:
Inclusion Criteria:

- All patients, whether adults or minors accompanied by their legal representative, who consulted in the orthodontics unit, and had access to the internet.

Exclusion Criteria:

- All patients who declined to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients present in the waiting room during the period of questionnaire distribution at the Orthodontic Unit of the Nice University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
online research of orthodontic information | At the inclusion
  Yes (score = 1) No (score = 2)

SECONDARY OUTCOMES:
trust in the information gathered | At the inclusion
  No confidence (score = 0) Moderate confidence (score = 1) Full confidence (score = 2)
The impact of online and social media information on orthodontic patients' decision-making | At the inclusion
  No influence (score = 0) Influenced decision (score = 1)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes-Maritimes, France